CLINICAL TRIAL: NCT07360171
Title: Validity Assessment of Sensors for Movement Tracking With Children/Youth With Diverse Neuromotor Abilities
Acronym: MOCAP
Status: Not yet recruiting | Type: Observational
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 0551
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy; Cerebral Palsy (CP)
Keywords: Home-Based Rehabilitation; Interactive Video Game Therapy; Gamified Rehabilitation; Digital Therapeutics; Tele-Rehabilitation; Active Video Gaming; Motion Analysis
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Arm: Participants' sociodemographic data is collected prior to the active component of study session. During the active component, participants will play a collection on movement-based video games that target specific rehabilitation movements. While playing, participants' movements are captured using different technologies including 2D and 3D cameras and marker-based motion capture systems. The games will be played in a randomized order, and the motion data will be collected for the full duration. The participants will be able to rest as needed between each mini game. The overall active game play will be approximately 30 minutes with approximately 10 minutes of walking (3-8 passes on a 5m track for children who are able) and active range of movement measurements.
  Interventions: Device: Validity Assessment of Sensors for Movement Tracking With Children/Youth With Diverse Neuromotor Abilities

INTERVENTIONS:
Device: Validity Assessment of Sensors for Movement Tracking With Children/Youth With Diverse Neuromotor Abilities — Participants will play active video games by moving their bodies while their movements are tracked by different sensors.

SUMMARY:
The overall goal of this study is to establish the clinical utility and accuracy of markerless motion captures systems for tracking therapy exercises and movement during game play. Specific aims are:

1. To evaluate the accuracy of the kinematic metrics tracked by marker-less motion capture systems by comparing them to the gold standard marker-based Motion Analysis system.
2. To assess agreement between exercise repetition counts and clinical assessment scores determined from data collected by the markerless motion capture systems compared to the gold standard marker-based Motion Analysis system and a trained clinician.
3. To explore the extent to which kinematic metrics collected during gameplay (e.g. smoothness of movement, symmetry index) can discriminate different motor abilities.
4. To understand children's perspectives on motion capture video games in the context of rehabilitation.

Participants will:

Perform active range of motion of each joint (3 repetitions, outside of the game environment) and rehabilitative movements within games developed at Holland Bloorview that target anatomical movements (e.g. shoulder abduction/adduction, shoulder flexion/extension, elbow flexion/extension, lateral trunk lean, hip flexion/extension, knee flexion/extension, trunk flexion/extension)

Play each mini game until 10 repetitions are made regarding the game objective or 2-minutes of game play is reached.

DETAILED DESCRIPTION:
Problems in prenatal brain development or brain injury in infancy can cause cerebral palsy (CP), a non-progressive disorder associated with impaired movement, posture, and balance. CP is the most common motor disability in children affecting two to three children for every 1000 births.

Although CP is a permanent disability, occupational and physical therapy can be implemented to help improve motor function or manage the symptoms over time. However, access to these therapies can be limited by financial, time, and geographical constraints. This motivates interest in home-based rehabilitation programs. Several studies have evaluated the possibility of active video games (AVGs) to complement conventional in-person rehabilitation interventions and boost motivation in children. The user interacts with the environment within the AVG via different motion-tracking interfaces ranging in complexity from inertial measurement units (i.e. Wii control stick) to 3D depth sensors (i.e. Microsoft Kinect). From a meta-analysis conducted by Ren et al., AVGs have been found to enhance gross motor function for children with CP.

Given the individual rehabilitation goals and abilities of each child, AVGs are most effective when they can be calibrated to target specific body segments for motor skill development. Ideally, AVGs would adapt to the child's physical performance in the same way that a therapist observes a patient's progress and adjusts the intensity and frequency of the exercise. Data collected from technological systems, such as an optoelectronic motion tracking system, has the potential to follow changes in movement abilities to support progress tracking. Gold standard optoelectronic motion capture (e.g., Vicon, Motion Analysis) are too expensive for the home, but there are low-cost, commercial products that are practical for home use (e.g., Microsoft Kinect, Orbbec Persee). While the movement-tracking capabilities of these devices are sufficient to support game play, it is not known how accurately they track movements (i) during game play and (ii) for children with diverse motor skills and patterns. This information is pertinent to validate the use of low-cost optoelectronic, motion-tracking to (i) provide high quality feedback and support practice of therapy exercises (e.g. to what extent can these systems recognize and provide feedback on exercises in the same way that a therapist would?) and (2) track changes in motor performance (i.e. to what extent can these systems be used to accurately quantify and track changes in motor skills?)

To increase accessibility for a larger population of children with CP, a series of interactive video games have been created at the Possibility Engineering and Research Lab (PEARL), which tracks rehabilitation exercises and integrates these into gameplay. The video games, Bootle Blast (BB) and Bootle Boot Camp (BC), utilize a 3D depth sensor, the Orbbec Persee+. Bootle Blast has been successfully piloted by 4 children with CP over 12 weeks in their homes and used in clinics at Holland Bloorview Kids Rehabilitation Hospital since 2017. To date, body tracking has been used primarily to support children's interactions in the games. Its accuracy for tracking therapy exercises, potential to deliver high quality feedback, and validity for quantifying qualities of movement (e.g., reach envelope, smoothness of movement, movement trajectory) has yet to be established.

The overall goal of this study is to establish the clinical utility and accuracy of markerless motion captures systems (e.g. the Orbbec Persee+/Astra 2, Apple LiDAR, 2D cameras + body tracking software) for tracking therapy exercises and movement during game play.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 5 to 24 years
2. Sufficient motor skills to successfully play the game (i.e., able to lift hand above shoulder)
3. Able to see and interact with the monitor - minimal visual or auditory impairments
4. Willing to wear reflective stickers on skin and on tight fitting clothing
5. Willing to wear athletic tape around arms and/or legs to secure loose clothing
6. Mobility similar to GMFCS Levels I-III.

Exclusion Criteria:

* Any injury/disability that would make moderate exercise unsafe.
* History of epilepsy aggravated by screen time. For the latter, the child will be eligible to participate if they safely participated in 1 hour of TV/video games per week as reported by the parent.

Ages: 5 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study population will include clients recruited through Holland Bloorview Kids Rehabilitation Hospital as well as through community postings
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized Clinical Assessment: 30 Second Sit To Stand Test | Baseline
  A measurement that assesses functional lower extremity strength.
Standardized Clinical Assessment - Five Times Sit to Stand Test | Baseline
  The Five Times Sit to Stand Test measures one aspect of transfer skill. The test provides a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements.
Standardized Clinical Assessment: Paediatric Reach Test | Baseline
  A modified form of the Functional Reach Test (FRT). The PRT measures side reaching as well as forward reaching in both sitting and standing positions.
Standardized Clinical Assessment: Single Leg Stance Test | Baseline
  Used to assess static postural and balance control
Standardized Clinical Assessment: Timed Up and Go | Baseline
  Assesses mobility, balance, walking ability, and fall risk
Sensor Movement Tracking Data | Baseline
  Joint positions in X-Y-Z coordinate space.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Biddiss, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital, Bloorview Research Institute
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No